CLINICAL TRIAL: NCT01245764
Title: Evaluation of Safety and Immunogenicity of GARDASIL™ in Healthy Females Between 9 and 26 Years of Age in SubSaharan Africa
Brief Title: GARDASIL™ Study in Healthy Females Between 9 and 26 Years of Age in Sub-Saharan Africa (V501-046)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V501-046
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Papillomavirus Infections
Keywords: Cervical cancer; vulvar cancer; vaginal cancer; genital warts; human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata | interventions — Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GARDASIL™ 9 to 12 Years Old (Experimental): GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Participants will not continue to study Phase B.
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)
- GARDASIL™ 13 to 15 Years Old (Experimental): GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Participants will not continue to study Phase B.
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)
- GARDASIL™ 16 to 26 Years Old (Experimental): GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Participants will not continue to study Phase B.
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)
- Placebo 9 to 12 Years Old (Placebo Comparator): Placebo to GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. After database lock and unblinding for study Phase A, participants will have the option to receive GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase B.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)
  Arms: GARDASIL™ 13 to 15 Years Old; GARDASIL™ 16 to 26 Years Old; GARDASIL™ 9 to 12 Years Old
Biological: Placebo
  Arms: Placebo 9 to 12 Years Old

SUMMARY:
The study is designed to determine the safety, tolerability and immunogenicity of a 3-dose regimen of GARDASIL™ administered to healthy females between 9 and 26 years of age, in Sub-Saharan Africa. Data from the current study are needed in order to complement existing extensive safety data from the GARDASIL™ clinical trials program, and confirm that GARDASIL™ may be administered safely and will induce immune responses in populations from and living in Sub-Saharan Africa, as GARDASIL™ has not previously been studied in this region of the world.

DETAILED DESCRIPTION:
In Phase A of the study, healthy females between 9 and 12 years of age will be randomized (4:1) to receive the 3-dose regimen of GARDASIL™ or placebo, and those between 13 and 26 years old will receive GARDASIL™. In Phase B of the study, participants who received placebo in Phase A will have the option to receive the 3-dose regimen of GARDASIL™.

ELIGIBILITY:
Inclusion Criteria :

* Healthy subjects who are native to and living in a participating Sub-Saharan African country.
* Subject agrees to provide study personnel with a primary telephone number as well as an alternate telephone number for follow-up purposes. If potential subject does not have a telephone number, the subject must provide an address at which he or she may be contacted.
* Post-pubertal female subjects must not be pregnant
* Subjects who are sexually active must agree to use effective contraception or remain abstinent through Month 7 of the study.
* Subjects who have not yet had sexual intercourse must either agree to remain abstinent through Month 7 of the study, or if they become sexually active during the vaccination phase of the study, to use effective contraception through Month 7.
* Subjects who have had sexual intercourse in the two weeks prior to enrollment must have been using effective contraception as defined above. (Emergency contraception is not considered effective contraception for enrollment in the study.)

Exclusion Criteria :

* Subject is pregnant as determined by a positive pregnancy test
* Subject has had a temperature ≥ 37.8 °C or ≥ 100 °F within 24 hours prior to the first injection.
* Subject is currently enrolled in another clinical study of an investigational agent or agents.
* Subject has a history of known prior vaccination with a HPV vaccine, or was previously enrolled in an HPV vaccine study and received either active agent or placebo.
* Subject has received any inactivated vaccine within 14 days prior to enrollment or any live vaccine within 21 days prior to enrollment.
* Subject has a history of severe allergic reaction to any agent (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention.
* Subject has known allergy to any vaccine component, including aluminum, yeast or BENZONASE™ (nuclease, Nycomed™ [used to remove residual nucleic acids from this and other vaccines]).
* Subject has received any immune globulin preparation or blood-derived products within the 6 months prior to the first injection, or plans to receive any such products during the course of the study.
* Subject has a history of splenectomy, known autoimmune disorder (e.g., systemic lupus erythematosus, rheumatoid arthritis), or is receiving immunosuppressives (e.g., substances or treatments known to diminish immune response such as radiation therapy, administration of antimetabolites, antilymphocytic sera, systemic corticosteroids). Individuals who have received periodic treatments with immunosuppressives, defined as at least 3 courses of systemic corticosteroids each lasting at least 1 week in duration for the year prior to enrollment, will be excluded. Subjects using topical steroids (i.e., inhaled or nasal) will be eligible for vaccination.
* Subject is immunocompromised or has been diagnosed as having Human Immunodeficiency Virus (HIV) infection
* Subject has known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Subject has known sickle cell anemia disease, active malaria or active tuberculosis.
* Subject has any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives.
* Subject has a history of recent or ongoing alcohol or other drug abuse.
* Female subject has a prior history of abnormal Pap test showing squamous intraepithelial lesion (SIL), atypical squamous cells of undetermined significance (ASC-US), atypical squamous cells, cannot rule out a high grade lesion (ASC-H), or biopsy showing cervical intraepithelial neoplasia (CIN) or worse.
* Subject has any prior history (or at Day 1) of genital warts or treatment for genital warts.
* Subject with >4 lifetime sexual partners.
* Subject has undergone hysterectomy with removal of the cervix.
* Subject plans to permanently relocate from the area prior to the completion of the study or to leave for an extended period of time when study visits would need to be scheduled.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2011-03-21 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mugo N, Ansah NA, Marino D, Saah A, Garner EI. Evaluation of safety and immunogenicity of a quadrivalent human papillomavirus vaccine in healthy females between 9 and 26 years of age in Sub-Saharan Africa. Hum Vaccin Immunother. 2015;11(6):1323-30. doi: 10.1080/21645515.2015.1008877. PMID 25912475
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V501-046&kw=V501-046&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- GARDASIL 9 to 12 Years Old; GARDASIL 13 to 15 Years Old; GARDASIL 16 to 26 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Immunogenicity was assessed at Month 7 of study Phase A and safety evaluation continued to Month 12 (total study duration up to 12 months). Participants did not continue to study Phase B.
- Placebo 9 to 12 Years Old: Placebo to GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Immunogenicity was assessed at Month 7 of study Phase A. After database lock and unblinding for study Phase A, participants had the option to receive GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase B. Safety evaluation continued to Month 7 of study Phase B (total study duration up to 19 months)
Period: Study Phase A
Arm/Group | GARDASIL 9 to 12 Years Old | GARDASIL 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Started | 80 | 30 | 120 | 20
Completed Vaccinations in Study Phase A | 77 | 28 | 117 | 19
Completed | 71 | 25 | 110 | 17
Not Completed | 9 | 5 | 10 | 3
Not completed — Other | 3 | 2 | 3 | 1
Not completed — Protocol Violation | 6 | 3 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 5 | 0
Period: Study Phase B
Arm/Group | GARDASIL 9 to 12 Years Old | GARDASIL 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Started | 0 | 0 | 0 | 17
Completed Vaccinations in Study Phase B | 0 | 0 | 0 | 17
Completed | 0 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GARDASIL 9 to 12 Years Old | GARDASIL 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old | Total
Number analyzed (Participants) | 80 | 30 | 120 | 20 | 250
Age, Customized [Number; unit: Participants]
  <9 years | 0 | 0 | 0 | 0 | 0
  9 to 12 years | 80 | 0 | 0 | 20 | 100
  13 to 15 years | 0 | 30 | 0 | 0 | 30
  16 to 26 years | 0 | 0 | 120 | 0 | 120
  >26 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 30 | 120 | 20 | 250
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 80 | 30 | 119 | 20 | 249
  Native Hawaiian or Other Pacific Island | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Seroconvert to Human Papillomavirus (HPV) Type 6
Description: Seroconversion was defined as achieving an anti-HPV Type 6 competitive Luminex Immunoassay (cLIA) level of >=20 milli Merck U/mL. The dilution-corrected limit of detection for the Type 6 cLIA was 4.2 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: Participants analyzed included those who received all 3 vaccinations in study Phase A and provided a sample for Month 7 serology testing. This analysis pooled results for participants receiving GARDASIL and compared these with results for participants receiving placebo.
Measure: Number; unit: Participants
Groups:
- GARDASIL 9 to 26 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A.
- Placebo 9 to 12 Years Old: Placebo to GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A.
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 147 | 13
Participants | 147 | 1

2. Primary Outcome: Number of Participants Who Seroconvert to HPV Type 11
Description: Seroconversion was defined as achieving an anti-HPV Type 11 cLIA level of >=16 milli Merck U/mL. The dilution-corrected limit of detection for the Type 11 cLIA was 3.9 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 147 | 13
Participants | 147 | 1

3. Primary Outcome: Number of Participants Who Seroconvert to HPV Type 16
Description: Seroconversion was defined as achieving an anti-HPV Type 16 cLIA level of >=20 milli Merck U/mL. The dilution-corrected limit of detection for the Type 16 cLIA was 9.7 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 160 | 14
Participants | 160 | 0

4. Primary Outcome: Number of Participants Who Seroconvert to HPV Type 18
Description: Seroconversion was defined as achieving an anti-HPV Type 18 cLIA level of >=24 milli Merck U/mL. The dilution-corrected limit of detection for the Type 18 cLIA was 5.8 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 156 | 14
Participants | 156 | 0

5. Primary Outcome: Number of Participants With Injection-site Adverse Experiences
Description: Participants were prompted to report injection-site experiences of pain, erythema, or swelling and were also asked to report any other injection-site adverse experiences
Time Frame: Up to Day 5 after any vaccination in study Phase A
Population: The analysis included all participants receiving at least 1 vaccination in study Phase A and who had postvaccination follow-up
Measure: Number; unit: Participants
Groups:
- GARDASIL 9 to 12 Years Old; Placebo 13 to 15 Years Old; GARDASIL 16 to 26 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A
- Placebo 9 to 12 Years Old: Placebo to match GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A
Arm/Group | GARDASIL 9 to 12 Years Old | Placebo 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 79 | 29 | 119 | 19
Participants | 54 | 21 | 88 | 9

6. Primary Outcome: Number of Participants With Elevated Temperature (Oral Temperature >=100 °F)
Time Frame: Up to Day 5 after any vaccination in study Phase A
Population: The analysis included all participants receiving at least 1 vaccination in study Phase A and who had temperature data
Measure: Number; unit: Participants
Arm/Group | GARDASIL 9 to 12 Years Old | Placebo 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 79 | 29 | 119 | 19
Participants | 9 | 6 | 7 | 5

7. Primary Outcome: Number of Participants With Serious Adverse Experiences
Description: A serious adverse experience is any adverse experience that results in death, is life threatening, results in persistent or significant disability/incapacity, results in or prolongs existing inpatient hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is another important medical event that may jeopardize the participant and may require medical or surgical intervention
Time Frame: From the time of informed consent is signed through the last study visit (up to 19 months)
Population: The analysis included all participants receiving at least 1 vaccination in study Phase A or B and who had postvaccination follow-up
Measure: Number; unit: Participants
Groups:
- Placebo 13 to 15 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Immunogenicity was assessed at Month 7 of study Phase A and safety evaluation continued to Month 12 (total study duration up to 12 months). Participants did not continue to study Phase B.
- GARDASIL 16 to 26 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Immunogenicity was assessed at Month 7 of study Phase A and safety evaluation will continue to Month 12 (total study duration up to 12 months). Participants did not continue to study Phase B.
Arm/Group | GARDASIL 9 to 12 Years Old | Placebo 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 79 | 29 | 119 | 19
Participants | 0 | 0 | 1 | 0

8. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-HPV Type 6 Antibody
Description: Anti-HPV Type 6 antibodies were measured by cLIA. The seropositive cut-off threshold for this assay is defined as 20 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 147 | 13
milli Merck U/mL | 602 [526 to 689] | NA [NA to NA] — GMT value was <10 milli Merck U/mL

9. Secondary Outcome: GMT of Anti-HPV Type 11 Antibody
Description: Anti-HPV Type 11 antibodies were measured by cLIA. The seropositive cut-off threshold for this assay is defined as 16 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 147 | 13
milli Merck U/mL | 626 [545 to 718] | NA [NA to NA] — GMT value was <7 milli Merck U/mL

10. Secondary Outcome: GMT of Anti-HPV Type 16 Antibody
Description: Anti-HPV Type 16 antibodies were measured by cLIA. The seropositive cut-off threshold for this assay is defined as 20 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 160 | 14
milli Merck U/mL | 3786 [3360 to 4265] | NA [NA to NA] — GMT value was <9 milli Merck U/mL

11. Secondary Outcome: GMT of Anti-HPV Type 18 Antibody
Description: Anti-HPV Type 18 antibodies were measured by cLIA. The seropositive cut-off threshold for this assay is defined as 24 milli Merck U/mL.
Time Frame: Month 7 (1 month postdose 3 in study Phase A)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | GARDASIL 9 to 26 Years Old | Placebo 9 to 12 Years Old
Number analyzed (Participants) | 156 | 14
milli Merck U/mL | 811 [708 to 928] | NA [NA to NA] — GMT value was <15 milli Merck U/mL

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to 19 months from study start. Other adverse events were assessed up to 15 days after each vaccination in study Phase A.
Description: The analysis included all participants receiving at least one vaccination and had at least one postvaccination follow-up visit.
Groups:
- GARDASIL 9 to 12 Years Old; GARDASIL 13 to 15 Years Old; GARDASIL 16 to 26 Years Old: GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. Participants did not continue to study Phase B.
- Placebo 9 to 12 Years Old: Placebo to GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase A. After database lock and unblinding for study Phase A, participants had the option to receive GARDASIL™ 0.5 mL injection at the Day 1, Month 2, and Month 6 visits in study Phase B.
Arm/Group | GARDASIL 9 to 12 Years Old | GARDASIL 13 to 15 Years Old | GARDASIL 16 to 26 Years Old | Placebo 9 to 12 Years Old
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/29 | 1/119 | 0/19
Other Adverse Events (participants affected / at risk) | 61/79 | 22/29 | 103/119 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GARDASIL 9 to 12 Years Old (N=79) | GARDASIL 13 to 15 Years Old (N=29) | GARDASIL 16 to 26 Years Old (N=119) | Placebo 9 to 12 Years Old (N=19)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GARDASIL 9 to 12 Years Old (N=79) | GARDASIL 13 to 15 Years Old (N=29) | GARDASIL 16 to 26 Years Old (N=119) | Placebo 9 to 12 Years Old (N=19)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 2 (3) | 8 (8) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Injection site erythema (General disorders) | 8 (12) | 3 (4) | 15 (21) | 1 (1)
Injection site pain (General disorders) | 53 (113) | 20 (46) | 88 (188) | 9 (21)
Injection site swelling (General disorders) | 23 (37) | 8 (9) | 31 (48) | 4 (7)
Pyrexia (General disorders) | 9 (12) | 6 (7) | 9 (10) | 5 (8)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 2 (3) | 2 (2) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (2) | 13 (14) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 27 (37) | 12 (16) | 41 (58) | 5 (7)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 11 (16) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.